CLINICAL TRIAL: NCT04454372
Title: Clinical Characteristics and Outcomes of 187 Critically Ill Patients With COVID-19
Brief Title: Clinical Characteristics and Outcomes of 187 Critically Ill Patients With Coronavirus Disease 2019 (COVID-19)
Status: Completed | Type: Observational
Sponsor: Hospital Sao Domingos (Other)
Responsible Party: Principal Investigator, José Raimundo Araujo de Azevedo, Principal investigator, Hospital Sao Domingos
Other Study IDs: covid-19 ICU
Record Dates: First submitted 2020-06-29; First posted 2020-07-01 (Actual); Last update posted 2022-03-29 (Actual); Status verified 2022-03

CONDITIONS: COVID-19
Keywords: COVID-19; critically ill patients; outcomes; treatment
MeSH Terms: conditions — COVID-19 | interventions — Demography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: demographic and clinical data obtained from hospital's electronic medical record. — This retrospective observational study. . Demographic and severity data will include age, sex, SAPS 3 and SOFA scores at admission, nutritional risk determined by NRS-2002 and commodities. Clinical and laboratory data on arrival at the ICU including PaO2 / FIO2, blood count and PCR D-dimer, ferritin, fibrinogen, DHL. Drug interventions including use of hydroxychloroquine, corticosteroids, heparin, tocilizumab. Characteristics of invasive and non-invasive respiratory support, use of prone position and ECMO and vasoactive drugs. The main complications, acute kidney injury requiring renal replacement therapy, secondary infectious complications will be documented as well as the outcomes.

SUMMARY:
This case series describes the clinical characteristics, treatment and outcomes of patients with laboratory confirmed COVID-19 admitted to a 35 beds intensive care unit of a tertiary hospital in Northeast Brazil.

DETAILED DESCRIPTION:
This retrospective observational study will be carried out at Hospital São Domingos, state of Maranhao, Brasil. It is a tertiary hospital with 450 beds and six Intensive Care Units (ICU) with a total of 63 beds. With the admission of the first patients with Coronavirus Disease 2019 (COVID-19) as of March 20, we initially made available a 12 beds ICU exclusively for the treatment of patients with COVID-19. At the beginning of April, the number of beds was increased to 35 and, immediately afterwards, two semi-intensive units (16 and 21 beds) were created for patients in need of non-invasive respiratory support, with the 35 beds ICU 35 dedicated to receive only patients in need of high-level support (usually invasive mechanical ventilation) with or without other organ dysfunctions.

In the period from March 20 to June 15, 2020, 935 patients with confirmed diagnosis (RT-PCR) of COVID-19 were admitted to the hospital and 187 of them were treated in the ICU.

Data were obtained from the hospital's electronic medical record. Demographic and severity data included age, sex, Simplified Acute Physiology 3 (SAPS 3) and Sequential Organ Failure Assessment (SOFA) scores at admission, nutritional risk determined by Nutritional Risk Screening 2002 (NRS-2002) and commodities. Clinical and laboratory data on arrival at the ICU including Partial pressure of oxygen in arterial bood / Inspired fraction of oxygen (PaO2 / FIO2) complete blood count and PCR D-dimer, ferritin, fibrinogen and lactic acid dehydrogenasew (LDH). Drug interventions including use of hydroxychloroquine, corticosteroids, heparin, tocilizumab. Characteristics of invasive and non-invasive respiratory support, use of prone position, ECMO and vasoactive drugs. The main complications, acute kidney injury requiring hemodialysis, secondary infectious complications will be documented as well as the outcomes.

ELIGIBILITY:
Inclusion Criteria:

* All patients admitted to the 35 beds ICU between March 20 and June 15, 2020 with laboratory confirmed diagnosis of COVID-19 (RT-PCR).

Exclusion Criteria:

* Patients admitted to the ICU in which the RT-PCR was negative, and patients that did not require high level life support (RRT, Prone position, ECMO, hemodymnamic monitoring and support).

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All critically ill patients admitted to the 35 beds ICU dedicated to COVID-19 in the period of March 20 and June 15, 2020 with laboratory confirmed diagnosis of COVID-19. Patients that could be managed without invasive mechanical ventilation and that did not require other high level life support were managed in one of the semi intensive units (16 and 21 beds).
Sampling Method: Probability Sample
Enrollment: 187 (Actual)
Dates: Start 2020-07-15 (Actual); Primary Completion 2020-09-20 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
Outcome 30 days after ICU admission | 30 days after admission
  A seven-category ordinal scale consisting of: 1. Death; 2. hospitalized, on invasive mechanical ventilation; 3. hospitalized, on non-invasive ventilation; 4. hospitalized, requiring supplemental oxygen; 5. hospitalized not requiring supplemental oxygen; 6. hospitalized, not requiring supplemental oxygen - no longer requires ongoing medical care. 7 Not hospitalized

CONTACTS AND LOCATIONS:
Overall Officials: JOSE AZEVEDO, MD, Study Chair — Hospital Sao Domingos
Locations (1):
- Hospital Sao Domingos, São Luís, Maranhão, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yang P, Tekwani S, Martin GS. In COVID-19, adding lopinavir-ritonavir to usual care did not shorten time to clinical improvement. Ann Intern Med. 2020 Jun 16;172(12):JC63. doi: 10.7326/ACPJ202006160-063. PMID 32539520
- [Background] Grein J, Ohmagari N, Shin D, Diaz G, Asperges E, Castagna A, Feldt T, Green G, Green ML, Lescure FX, Nicastri E, Oda R, Yo K, Quiros-Roldan E, Studemeister A, Redinski J, Ahmed S, Bernett J, Chelliah D, Chen D, Chihara S, Cohen SH, Cunningham J, D'Arminio Monforte A, Ismail S, Kato H, Lapadula G, L'Her E, Maeno T, Majumder S, Massari M, Mora-Rillo M, Mutoh Y, Nguyen D, Verweij E, Zoufaly A, Osinusi AO, DeZure A, Zhao Y, Zhong L, Chokkalingam A, Elboudwarej E, Telep L, Timbs L, Henne I, Sellers S, Cao H, Tan SK, Winterbourne L, Desai P, Mera R, Gaggar A, Myers RP, Brainard DM, Childs R, Flanigan T. Compassionate Use of Remdesivir for Patients with Severe Covid-19. N Engl J Med. 2020 Jun 11;382(24):2327-2336. doi: 10.1056/NEJMoa2007016. Epub 2020 Apr 10. PMID 32275812
- [Background] Alhazzani W, Moller MH, Arabi YM, Loeb M, Gong MN, Fan E, Oczkowski S, Levy MM, Derde L, Dzierba A, Du B, Aboodi M, Wunsch H, Cecconi M, Koh Y, Chertow DS, Maitland K, Alshamsi F, Belley-Cote E, Greco M, Laundy M, Morgan JS, Kesecioglu J, McGeer A, Mermel L, Mammen MJ, Alexander PE, Arrington A, Centofanti JE, Citerio G, Baw B, Memish ZA, Hammond N, Hayden FG, Evans L, Rhodes A. Surviving Sepsis Campaign: guidelines on the management of critically ill adults with Coronavirus Disease 2019 (COVID-19). Intensive Care Med. 2020 May;46(5):854-887. doi: 10.1007/s00134-020-06022-5. Epub 2020 Mar 28. PMID 32222812
- [Result] Guan WJ, Ni ZY, Hu Y, Liang WH, Ou CQ, He JX, Liu L, Shan H, Lei CL, Hui DSC, Du B, Li LJ, Zeng G, Yuen KY, Chen RC, Tang CL, Wang T, Chen PY, Xiang J, Li SY, Wang JL, Liang ZJ, Peng YX, Wei L, Liu Y, Hu YH, Peng P, Wang JM, Liu JY, Chen Z, Li G, Zheng ZJ, Qiu SQ, Luo J, Ye CJ, Zhu SY, Zhong NS; China Medical Treatment Expert Group for Covid-19. Clinical Characteristics of Coronavirus Disease 2019 in China. N Engl J Med. 2020 Apr 30;382(18):1708-1720. doi: 10.1056/NEJMoa2002032. Epub 2020 Feb 28. PMID 32109013
- [Result] Richardson S, Hirsch JS, Narasimhan M, Crawford JM, McGinn T, Davidson KW; the Northwell COVID-19 Research Consortium; Barnaby DP, Becker LB, Chelico JD, Cohen SL, Cookingham J, Coppa K, Diefenbach MA, Dominello AJ, Duer-Hefele J, Falzon L, Gitlin J, Hajizadeh N, Harvin TG, Hirschwerk DA, Kim EJ, Kozel ZM, Marrast LM, Mogavero JN, Osorio GA, Qiu M, Zanos TP. Presenting Characteristics, Comorbidities, and Outcomes Among 5700 Patients Hospitalized With COVID-19 in the New York City Area. JAMA. 2020 May 26;323(20):2052-2059. doi: 10.1001/jama.2020.6775. PMID 32320003
- [Result] Zhang C, Wu Z, Li JW, Zhao H, Wang GQ. Cytokine release syndrome in severe COVID-19: interleukin-6 receptor antagonist tocilizumab may be the key to reduce mortality. Int J Antimicrob Agents. 2020 May;55(5):105954. doi: 10.1016/j.ijantimicag.2020.105954. Epub 2020 Mar 29. PMID 32234467
- [Result] Mehta P, McAuley DF, Brown M, Sanchez E, Tattersall RS, Manson JJ; HLH Across Speciality Collaboration, UK. COVID-19: consider cytokine storm syndromes and immunosuppression. Lancet. 2020 Mar 28;395(10229):1033-1034. doi: 10.1016/S0140-6736(20)30628-0. Epub 2020 Mar 16. No abstract available. PMID 32192578
- [Result] Wu C, Chen X, Cai Y, Xia J, Zhou X, Xu S, Huang H, Zhang L, Zhou X, Du C, Zhang Y, Song J, Wang S, Chao Y, Yang Z, Xu J, Zhou X, Chen D, Xiong W, Xu L, Zhou F, Jiang J, Bai C, Zheng J, Song Y. Risk Factors Associated With Acute Respiratory Distress Syndrome and Death in Patients With Coronavirus Disease 2019 Pneumonia in Wuhan, China. JAMA Intern Med. 2020 Jul 1;180(7):934-943. doi: 10.1001/jamainternmed.2020.0994. PMID 32167524